CLINICAL TRIAL: NCT01120145
Title: Assessment of the Efficacy and Effectiveness of Sulphadoxine-pyrimethamine for Intermittent Preventive Treatment of Malaria in Pregnancy in Malawi
Brief Title: Assessment of Sulphadoxine-pyrimethamine for Intermittent Preventive Treatment of Malaria in Pregnancy in Malawi
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Kamuzu University of Health Sciences (Other)
Responsible Party: Jacek Skarbinski, Malaria Branch, Centers for Disease Control and Prevention
Other Study IDs: CDC-CGH-5756
Record Dates: First submitted 2010-05-05; First posted 2010-05-10 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Malaria in Pregnancy
Keywords: Malaria; Pregnancy; Sulphadoxine-pyrimethamine
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Blood spots will be collected from parasitemic patients to look at malaria prasite molecular markers of resistance to sulphadoxine-pyrimethamine.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Therapeutic efficacy study: Asymptomatic parasitemic pregnant women at 16-26 weeks of gestation will be enrolled into the study and followed weekly for 42 days after the receipt of sulphadoxine-pyrimethamine intermittent preventive treatment in pregnancy to assess the clearance of parasitemia.
- Birth outcomes study: Women presenting for delivery will be enrolled and assessed for a history of sulphadoxine-pyrimethamine intermittent preventive treatment in pregnancy and evidence of malaria infection by placental histology, maternal peripheral parasitemia, maternal anemia and infant cord blood parasitemia.
- Characterizing molecular markers of SP resistance: Parasitemic outpatients attending the health facility will be tested for parasite molecular markers of sulphadoxine-pyrimethamine resistance.

SUMMARY:
The purpose of this study is to determine the efficacy and effectiveness of sulphadoxine-pyrimethamine intermittent preventive treatment in pregnancy for reducing malaria-associated morbidity in pregnant women in Malawi.

DETAILED DESCRIPTION:
Malaria infection in pregnancy is associated with severe maternal anemia, placental parasitemia, low birth weight, and increased perinatal mortality. Intermittent preventive treatment in pregnancy (IPTp) with sulphadoxine-pyrimethamine (SP) is recommended by the World Health Organization (WHO) for reducing the risks associated with malaria in pregnancy. Traditionally, the level of SP resistance has been assessed by monitoring its in vivo efficacy for treatment of uncomplicated malaria in children under five years of age. However, parasite resistance to SP has compromised its efficacy in young children, and SP is no the longer a first-line recommended treatment for malaria in most African countries. Although SP currently appears to remain effective for IPTp in pregnant women probably because they have more immunity than young children, it is important to monitor SP effectiveness in this population. Characterizing SP resistance through in vivo and molecular methods in pregnant women may be useful to predict whether to continue a policy of IPTp with SP.

There will be three parts to this study. To determine therapeutic efficacy of SP IPTp in pregnant women, a prospective in vivo study will be done in women who present for antenatal care (ANC). Women will receive SP IPTp according to national guidelines and will be followed for 42 days for clearance of peripheral parasitemia. To determine birth outcomes of women given SP IPTp, a retrospective cohort study will be performed assessing outcomes of women at delivery. Information on prior receipt of SP IPTp, peripheral and placental parasitemia at delivery, placental histology, maternal anemia, and birth weight will be collected. To characterize baseline resistance of SP in pregnant women and in the general population, parasites will be collected from both participating women and attendees at outpatient clinics to measure SP resistance markers.

The results of this study will be used by the Malawi national control program to evaluate current policy of using SP for IPTp. This study will also contribute towards an international effort led by WHO to align priorities and methodologies in gathering data on the efficacy of SP in IPTp in the face of increasing SP resistance, thus providing data to inform IPTp policy at the global level.

ELIGIBILITY:
Therapeutic efficacy study

Inclusion Criteria:

* 16-26 weeks gestation based on last menstrual period (LMP) or quickening
* Axillary temperature <37.5 degrees Celsius
* Informed consent

Exclusion Criteria:

* History of hypersensitivity reaction to SP or components of SP
* Axillary temperature ≥37.5 degrees C
* History of receipt of antimalarials in the past month
* Known HIV infection

Birth outcomes study:

Inclusion Criteria:

* Singleton pregnancy
* SP IPTp history available
* Informed consent

Exclusion Criteria:

* Blood transfusion after the 16th gestational week
* Receipt of antimalarials other than SP for IPTp after 16th gestational week
* Known HIV infection

Characterizing molecular markers of SP resistance:

Inclusion Criteria:

* Outpatient attending selected health facility
* Informed consent

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Therapeutic efficacy study: Asymptomatic parasitemic pregnant women at 16-26 weeks of gestation Birth outcomes study: Pregnant women presenting for delivery Characterizing molecular markers of SP resistance study: Parasitemic outpatients
Sampling Method: Non-Probability Sample
Enrollment: 1410 (Actual)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Therapeutic efficacy study: Development of fever or symptoms of severe malaria (defined by WHO) and parasitemia at any time after the first dose of SP during the 42 day follow up period | 42 days
Birth outcomes study: Evidence of malaria infection based on placental histology at the time of delivery | At time of birth
Characterizing molecular markers of SP resistance: Prevalence of molecular markers of sulphadoxine-pyrimethamine resistance at the time of health facility visit | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Skarbinski, MD, Principal Investigator — Malaria Branch, Centers for Disease Control and Prevention; Don Mathanga, MD, PhD, Principal Investigator — Kamuzu University of Health Sciences
Locations (1):
- Machinga District Hospital, Liwonde, Machinga District, Malawi

REFERENCES:
- [Derived] Gutman J, Mwandama D, Wiegand RE, Abdallah J, Iriemenam NC, Shi YP, Mathanga DP, Skarbinski J. In vivo efficacy of sulphadoxine-pyrimethamine for the treatment of asymptomatic parasitaemia in pregnant women in Machinga District, Malawi. Malar J. 2015 May 13;14:197. doi: 10.1186/s12936-015-0710-7. PMID 25962439